CLINICAL TRIAL: NCT06308718
Title: A Long-term Follow-up Study to Evaluate Safety and Efficacy of Krabbe Patients From Gene Therapy Clinical Trials Involving the Administration of FBX-101 (AAVrh.10-hGALC)
Brief Title: Long-term Follow-up Study to Evaluate Safety and Efficacy of FBX-101 in Krabbe Patients
Status: Terminated | Type: Observational
Why Stopped: The FBX-101 clinical program has been discontinued by Forge Biologics
Sponsor: Forge Biologics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: FBX-101-LTFU
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Krabbe Disease
Keywords: Lysosomal Storage Disorder; Globoid Cell Leukodystrophy; Leukodystrophy; GALC
MeSH Terms: conditions — Leukodystrophy, Globoid Cell; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Peripheral Blood Mononuclear Cells, Plasma, Urine, Faces, Saliva.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled in the FBX-101-LTFU study: The participants will be followed for 36 months after they have concluded their participation in the interventional trial. They will complete 5 scheduled visits with assessments as specified in the schedule of assessments, to collect data for safety and additional signs of efficacy for FBX-101. Those patients enrolled from any other early terminated trial, will first complete pending evaluations from that trial.
  Interventions: Biological: FBX-101

INTERVENTIONS:
Biological: FBX-101 — A replication-deficient adeno-associated virus gene transfer vector expressing the human galactocerebrosidase (hGALC) cDNA will be delivered one-time through a venous catheter inserted into a peripheral limb vein.

SUMMARY:
This is an observational study that will enroll any patients with Krabbe disease that have participated in prior interventional clinical trials involving the administration of FBX-101.

DETAILED DESCRIPTION:
FBX-101-LTFU is a multicenter, non-interventional, Long-Term Follow-Up (LTFU) study of participants from prior interventional trials involving the administration of FBX-101. Eligible participants will undergo clinical evaluations at prespecified intervals for at least 3 years from the last visit in the prior clinical trial (up to 5 years post-FBX-101 treatment). Overall safety and additional signs of efficacy will be collected with a series of laboratory tests, diagnostic tests, and performance surveys. Additionally, children participating in interventional trials that are terminated early will be transferred to this LTFU study and will complete any pending visits from the interventional trial before starting the clinical evaluations included in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participants that have completed a prior clinical trial involving the administration of FBX-101.
* Parent(s)/legal guardian(s) of participant willing and able to complete the informed consent process and comply with study procedures and visit schedule.

Exclusion Criteria:

•Planned or current participation in any other interventional clinical study that may confound the safety or efficacy evaluation of FBX-101 during this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is an observational long-term follow-up (LTFU) study of participants from prior interventional trials involving the administration of FBX-101.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Long Term safety as assessed by incidence of Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) that are attributed to FBX-101 | 36 months

SECONDARY OUTCOMES:
Efficacy as assessed by change of gross motor function measured longitudinally by Peabody Developmental Motor Scale (PDMS-2) | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of gross motor function measured longitudinally by Bruininks-Oseretsky Test of Motor Proficiency (BOT-2) | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of gross motor function measured longitudinally by Gross Motor Function Measure 88 (GMFM-88) | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of fine motor function measured longitudinally by Mullen Scales of Early Learning (MSEL) | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of fine motor function measured longitudinally by Beery VMI Sixth Edition (VMI) | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of fine motor function measured longitudinally by Bayley Scales of Infant Development (Bayley-III) | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of fine motor function measured longitudinally by Vineland Adaptive Behavior Scale (Vineland 3) | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of cognitive function measured longitudinally by Mullen Scales of Early Learning (MSEL) | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of cognitive function measured longitudinally by the Differential Ability Scale II (DAS-II) | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of cognitive function measured longitudinally by Bayley Scales of Infant Development (Bayley-III) | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of adaptive behaviour function measured longitudinally by Vineland Adaptive Behavior Scale (Vineland 3). | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of language function measured longitudinally by Mullen Scales of Early Learning (MSEL). | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of language function measured longitudinally by Clinical Evaluation of Language Fundamentals Fifth Edition (CELF-5) | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of language function measured longitudinally by Bayley Scales of Infant Development (Bayley-III) | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of language function measured longitudinally by Vineland Adaptive Behavior Scale (Vineland 3). | 36 months
  The site is providing raw data and sponsor is calculating derived scores according to specific manual. Higher values will mean better outcome.
Efficacy as assessed by change of quality of life measured longitudinally by the Pediatric Quality of Life (PedsQL) Generic Core Scales with Family Impact Module and Multidimensional Fatigue Scale | 36 months
Efficacy as assessed by change of developmental milestones such as language and motor skills as measured longitudinally by an specific Developmental Milestones questionnaire | 36 months
Efficacy as assessed by change of hearing function measured longitudinally by Auditory Brainstem Responses (ABRs) | 36 months
  Absolute values for Waves I, III and V in milliseconds will be recorded along interpretation and waveform morphology; and also Auditory Brainstem Responses (corrected).
Efficacy as assessed by change of hearing function measured longitudinally by Behavior Audiometry (BAUD) | 36 months
Efficacy as assessed by change of peripheral nerve conduction velocity measured longitudinally by Nerve Conduction Velocity (NCV) assessments | 36 months
Efficacy as assessed by change of Fractional Anisotropy (FA) as measured longitudinally by brain Magnetic Resonance Imaging (MRI) with Diffusion Tensor Imaging (DTI) | 36 months
Efficacy as assessed by change of visual function as measured longitudinally by visual evoked potentials (VEP) | 36 months
Efficacy as assessed by change of visual function as measured longitudinally by visual acuity | 36 months
Efficacy as assessed by change of whole blood donor chimerism | 36 months
Efficacy as assessed by change of psychosine in whole blood and plasma | 36 months
Efficacy as assessed by change of Galactosylceramidase (GALC) levels in plasma and Cerebrospinal Fluid (CSF) | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Hospitals - Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bascou N, DeRenzo A, Poe MD, Escolar ML. A prospective natural history study of Krabbe disease in a patient cohort with onset between 6 months and 3 years of life. Orphanet J Rare Dis. 2018 Aug 9;13(1):126. doi: 10.1186/s13023-018-0872-9. PMID 30089515
- [Background] Beltran-Quintero ML, Bascou NA, Poe MD, Wenger DA, Saavedra-Matiz CA, Nichols MJ, Escolar ML. Early progression of Krabbe disease in patients with symptom onset between 0 and 5 months. Orphanet J Rare Dis. 2019 Feb 18;14(1):46. doi: 10.1186/s13023-019-1018-4. PMID 30777126
- [Background] Escolar ML, Poe MD, Provenzale JM, Richards KC, Allison J, Wood S, Wenger DA, Pietryga D, Wall D, Champagne M, Morse R, Krivit W, Kurtzberg J. Transplantation of umbilical-cord blood in babies with infantile Krabbe's disease. N Engl J Med. 2005 May 19;352(20):2069-81. doi: 10.1056/NEJMoa042604. PMID 15901860
- [Background] Yoon IC, Bascou NA, Poe MD, Szabolcs P, Escolar ML. Long-term neurodevelopmental outcomes of hematopoietic stem cell transplantation for late-infantile Krabbe disease. Blood. 2021 Apr 1;137(13):1719-1730. doi: 10.1182/blood.2020005477. PMID 33150395
- [Background] Wright MD, Poe MD, DeRenzo A, Haldal S, Escolar ML. Developmental outcomes of cord blood transplantation for Krabbe disease: A 15-year study. Neurology. 2017 Sep 26;89(13):1365-1372. doi: 10.1212/WNL.0000000000004418. Epub 2017 Aug 30. PMID 28855403
- [Background] Gupta A, Poe MD, Styner MA, Panigrahy A, Escolar ML. Regional differences in fiber tractography predict neurodevelopmental outcomes in neonates with infantile Krabbe disease. Neuroimage Clin. 2014 Sep 26;7:792-8. doi: 10.1016/j.nicl.2014.09.014. eCollection 2015. PMID 25844309
- [Background] Bradbury AM, Bagel J, Swain G, Miyadera K, Pesayco JP, Assenmacher CA, Brisson B, Hendricks I, Wang XH, Herbst Z, Pyne N, Odonnell P, Shelton GD, Gelb M, Hackett N, Szabolcs P, Vite CH, Escolar M. Combination HSCT and intravenous AAV-mediated gene therapy in a canine model proves pivotal for translation of Krabbe disease therapy. Mol Ther. 2024 Jan 3;32(1):44-58. doi: 10.1016/j.ymthe.2023.11.014. Epub 2023 Nov 11. PMID 37952085
- [Background] Siddiqi ZA, Sanders DB, Massey JM. Peripheral neuropathy in Krabbe disease: effect of hematopoietic stem cell transplantation. Neurology. 2006 Jul 25;67(2):268-72. doi: 10.1212/01.wnl.0000230156.01228.33. PMID 16864820
- [Background] Vander Lugt MT, Chen X, Escolar ML, Carella BA, Barnum JL, Windreich RM, Hill MJ, Poe M, Marsh RA, Stanczak H, Stenger EO, Szabolcs P. Reduced-intensity single-unit unrelated cord blood transplant with optional immune boost for nonmalignant disorders. Blood Adv. 2020 Jul 14;4(13):3041-3052. doi: 10.1182/bloodadvances.2020001940. PMID 32634238